CLINICAL TRIAL: NCT01382160
Title: Serum Concentration of Adalimumab (Humira) as a Predictive Factor of Clinical Outcomes in Rheumatoid Arthritis (AFORA)
Brief Title: Serum Concentration of Adalimumab as a Predictive Factor of Clinical Outcomes in Rheumatoid Arthritis (AFORA)
Acronym: AFORA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHRI10-DM/AFORA; 2010-021449-28 (EudraCT Number); A100898-30 (Other: Afssaps); 2010-R24 (Other: CPP)
Record Dates: First submitted 2010-12-02; First posted 2011-06-27 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; adalimumab; pharmacokinetic-pharmacodynamic relationship; immunogenicity; Fc gamma receptors polymorphisms
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adalimumab (Experimental): 40 mg every two weeks, by subcutaneous way
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — 40 mg every two weeks, by subcutaneous way
  Other Names: Humira

SUMMARY:
Adalimumab is a fully human monoclonal antibody to tumor necrosis factor-alpha (TNF-α) approved in rheumatoid arthritis (RA) refractory to disease modifying anti rheumatic drugs (DMARDs) and for the treatment of severe, active and progressive RA in adults not previously treated with methotrexate.

However, almost one third of patients have no response and approximately 15% develop antibodies towards adalimumab (ATA) after a 6 month course of treatment. There is a relationship between adalimumab concentration and clinical response obtained after 6 month of treatment. Furthermore adalimumab concentration measured 3 months after initiation seems to predict the clinical response at 6 months.

There is an important inter individual pharmacokinetic variability of adalimumab. Side effects may occur at the recommended dose and more than 3 months of treatment are generally required to estimate the clinical response.

A therapeutic drug monitoring could help clinicians to early adjust the dose to optimize the response and to avoid dose related side effects. To date there is no definite adalimumab target concentration predictive of the clinical response to allow such a pharmacologic monitoring.

ELIGIBILITY:
Inclusion Criteria:

* RA according to the American College of Rheumatology (ACR) 1987 criteria
* Treatment with Adalimumab has been chosen by the physician / patient
* Treatment given in accordance to the SPC
* Stable Disease modifying anti rheumatic drugs (DMARDs) and glucocorticoids 4 weeks before enrollment and during the study period.
* Signed consent

Exclusion Criteria:

* more than one previous treatment with anti TNF-alpha
* Past history of malignancy, AIDS
* Pregnancy
* Change in DMARDS or glucocorticoid dose 4 weeks before entering the study
* Active or latent tuberculosis, other active infections
* Surgery scheduled during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To characterize the concentration-effect relationship of adalimumab in rheumatoid arthritis | During the 26 weeks of follow up.
  The primary objective is to characterize the concentration-effect relationship of adalimumab in rheumatoid arthritis (RA). To this aim, adalimumab concentration on the one hand and clinical and biological markers of disease activity on the other hand will be measured at baseline, week 4, week 8, week 12 and at week 26. Pharmacodynamic (PD) parameters will be estimated using PK(pharmacokinetic)-PD models in which Emax (maximum effect) and EC50 (concentration at which the effect is 50% of the maximum) will describe adalimumab effect on each markers of response.

SECONDARY OUTCOMES:
To study the relationship between genetic factors, immunogenicity and response to adalimumab in rheumatoid arthritis | During the 26 weeks of follow up.
  The secondary endpoints consist on the association study between FCGR3A polymorphisms, transcriptomic analysis (at baseline), presence of antibodies toward adalimumab (ATA) on the one hand and estimited individuals pharmacodynamic parameters on the other hand. Measurements will be carried out at baseline, week 4, week 8, week 12 and at week 26.

CONTACTS AND LOCATIONS:
Overall Officials: Denis MULLEMAN, MD, PhD, Principal Investigator — CHRU de Tours
Locations (7):
- France (7):
  - CHRU de Brest, Brest
  - CHR du Mans, Le Mans
  - CHRU de Nantes, Nantes
  - CHR d'Orléans, Orléans
  - CHRU de Poitiers, Poitiers
  - CHRU de Rennes, Rennes
  - CHRU de Tours, Tours

REFERENCES:
- [Result] Moulin D, Millard M, Taieb M, Michaudel C, Aucouturier A, Lefevre A, Bermudez-Humaran LG, Langella P, Sereme Y, Wanherdrick K, Gautam P, Mariette X, Dieude P, Gottenberg JE, Jouzeau JY, Skurnik D, Emond P, Mulleman D, Sellam J, Sokol H. Counteracting tryptophan metabolism alterations as a new therapeutic strategy for rheumatoid arthritis. Ann Rheum Dis. 2024 Feb 15;83(3):312-323. doi: 10.1136/ard-2023-224014. PMID 38049981